CLINICAL TRIAL: NCT01068210
Title: Lung Cancer Exercise Training Study: A Randomized Trial of Aerobic Training, Resistance Training, or Both in Lung Cancer Patients
Brief Title: Lung Cancer Exercise Training Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-215
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
Keywords: Exercise Intervention; Lung Cancer; 15-215
MeSH Terms: conditions — Lung Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aerobic Training (Experimental): A customized and supervised endurance exercise training program that will last 4 months (16 weeks). The regimen will be tailored to the individual fitness level. The exercise program will consist of three supervised sessions per week. During each session, the participant will cycle on a stationary bicycle at moderate intensity for approximately 30-60 minutes.
  Interventions: Behavioral: Aerobic Training
- Resistance Training (Experimental): A customized and supervised resistance exercise training program that will last 4 months (16 weeks). Resistance training will be performed on stationary weight machines, modification in equipment may be made by Exercise Physiologist. Patients will be progressively trained to perform two to three sets of 75-85% of maximal strength The participant will be trained to perform different resistance exercise, alternating between lower and upper body muscle groups. The exercise program will consist of three supervised sessions per week. Each session will last approximately 30-60 minutes.
  Interventions: Behavioral: Resistance Training
- Combined Aerobic and Resistance Training (Experimental): A customized and supervised endurance exercise training program that will last 4 months (16 weeks). The regimen will be tailored to the individual fitness level, and will be a combination of Arm A and Arm B, described above. At each session, the participant will complete aerobic training on a stationary bicycle and also resistance training using stationary weight machines. The exercise program will consist of three supervised sessions per week. Each session will last approximately 30-90 minutes.
  Interventions: Behavioral: Aerobic and Resistance Training
- Progressive Stretching Group (Attention-Control) (Active Comparator): A customized and supervised progressive stretching program that will last 4 months (16 weeks). The progressive stretching program will consist of a series of stretching exercises alternating between lower and upper body muscle groups/joints. This program will consist of three exercise sessions a week. Each session will last approximately 30-60 minutes.
  Interventions: Behavioral: Progressive Stretching

INTERVENTIONS:
Behavioral: Aerobic Training — The overall goal for all the exercise training groups will be 3 supervised exercise sessions per week an intensity between 50 to 100% of the individually determined VO2peak for aerobic training and an intensity between 50% to 85% of 1-RM for resistance training. All the exercise interventions are designed such that participants begin exercising at a low intensity (~50%-60% VO2peak / 1RM) that is subsequently increased to more moderate to vigorous intensity (~70%-100% VO2peak / ~70-85% 1RM) when appropriate. All interventions will be individually tailored to each patient following the principles of aerobic or resistance training prescription guidelines for adults.
  Arms: Aerobic Training
Behavioral: Progressive Stretching — The ultimate goal for the progressive stretching program is 3 individual stretching sessions. All sessions are required to be supervised. Duration of the stretching sessions is prescribed and implemented in accordance with standard stretching and flexibility training principles. This approach will be applied to guide each participant's prescribed stretching plan, with dose and scheduling modifications made by exercise physiologists, as required.
  Arms: Progressive Stretching Group (Attention-Control)
Behavioral: Resistance Training — The ultimate goal for resistance training alone is 3 resistance training session/week at an intensity above 50% to 85% of 1-RM for 30-60 minutes/session. Resistance trainings will be performed on stationary weight machines, modification in equipment may be made by Exercise Physiologist. Participants will be progressively trained to perform two to three sets of 75-85% of maximal strength.
  Arms: Resistance Training
Behavioral: Aerobic and Resistance Training — The ultimate goal will be three combined exercise sessions per week at an intensity above 50% VO2speak and above 50% 1-RM for aerobic and resistance training, respectively for 30-90 minutes/session.
  Arms: Combined Aerobic and Resistance Training

SUMMARY:
The purpose of the study is look at the effects of different types of exercise training with a stretching group and its effect on lung cancer patients. Subjects will take part in a 16 week training intervention that can consist of aerobic, resistance, aerobic & resistance, or a control group. Pre and Post testing will include stress tests, echos, blood, and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of study-related procedures
* Age 21 - 80 years
* Weight < 205 kgs
* ECOG ≤ 1
* Diagnosed with histologically confirmed lung cancer, regardless of disease stage and receiving any prior line of any therapy in the context of metastatic disease
* An interval of at least three months following the completion of primary resection, if appropriate
* An interval of no longer than ten years following completion of primary therapy, if appropriate
* Life expectancy ≥ 4 months
* Performing less than 150 minutes of structured moderate-intensity or strenuous-intensity exercise per week
* Exercise intolerance (i.e., patients must have a VO2peak below that predicted for active age and sex-matched individuals)
* Willing to be randomized to one of the study arms
* Willing to commit to the study program and comply with all related protocol procedures
* Able to achieve an acceptable peak baseline CPET, as defined by any of the following criteria:

  * achieving a plateau in oxygen consumption, concurrent with an increase in power output;
  * a respiratory exchange ratio ≥ 1.10;
  * attainment of maximal predicted heart rate (HRmax) (i.e., within 10 bpm of age-predicted HRmax [HRmax = 220-Age[years]);
  * volitional exhaustion, as measured by a rating of perceived exertion (RPE) ≥ 18 on the BORG scale.
* Able to complete an acceptable baseline CPET in the absence of high risk ECG findings or other inappropriate response to exercise as determined by the PI.
* Ability to achieve and complete an acceptable baseline one-repetition maximum muscular strength test as defined by the effective execution of protocol-specific joint and muscle ranges of motion without remarkable signs or symptoms of pain, discomfort or distress.

Exclusion Criteria:

* Presence of a concurrent, actively treated other malignancy, or history of other malignancy treated within the past 3 years (other than non-melanoma skin cancer);
* Room air desaturation at rest ≤ 85%;
* Mental impairment leading to inability to cooperate.
* Any of the following absolute contraindications to cardiopulmonary exercise testing:

  * Acute myocardial infarction (within 3-5 days of any planned study procedures);
  * Unstable angina;
  * Uncontrolled arrhythmia causing symptoms or hemodynamic compromise;
  * Recurrent syncope;
  * Active endocarditis;
  * Acute myocarditis or pericarditis;
  * Symptomatic severe aortic stenosis;
  * Uncontrolled heart failure;
  * Acute (within 3 months) pulmonary embolus or pulmonary infarction;
  * Thrombosis of lower extremities;
  * Suspected dissecting aneurysm;
  * Uncontrolled asthma;
  * Pulmonary edema;
  * Respiratory failure;
  * Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Jones, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Scott JM, Thomas SM, Herndon JE 2nd, Douglas PS, Yu AF, Rusch V, Huang J, Capaci C, Harrison JN, Stoeckel KJ, Nilsen T, Edvardsen E, Michalski MG, Eves ND, Jones LW. Effects and tolerability of exercise therapy modality on cardiorespiratory fitness in lung cancer: a randomized controlled trial. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1456-1465. doi: 10.1002/jcsm.12828. Epub 2021 Oct 17. PMID 34658160
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aerobic Training | Resistance Training | Combined Aerobic and Resistance Training | Progressive Stretching Group (Attention-Control)
Started | 24 | 23 | 20 | 23
Completed | 23 | 20 | 18 | 20
Not Completed | 1 | 3 | 2 | 3
Not completed — Lost to Follow-up | 1 | 2 | 2 | 1
Not completed — Second cancer | 0 | 1 | 0 | 0
Not completed — Disease progression | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Training | Resistance Training | Combined Aerobic and Resistance Training | Progressive Stretching Group (Attention-Control) | Total
Number analyzed (Participants) | 24 | 23 | 20 | 23 | 90
Age, Continuous [Mean (Full Range); unit: years] | 65 [44 to 76] | 64 [46 to 81] | 63 [32 to 78] | 67 [54 to 85] | 65 [32 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 13 | 16 | 59
  Male | 9 | 8 | 7 | 7 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 20 | 19 | 19 | 78
  Not Hispanic or Latino | 3 | 3 | 1 | 4 | 11
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 8 | 2 | 3 | 15
  White | 20 | 14 | 18 | 19 | 71
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 20 | 23 | 90

OUTCOME MEASURES:

1. Primary Outcome: Changes in VO2peak (on Exercise Capacity)
Description: To compare the efficacy of different types of exercise training modalities, relative to progressive stretching (attention control group)
Time Frame: 17 weeks
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Aerobic Training | Resistance Training | Combined Aerobic and Resistance Training | Progressive Stretching Group (Attention-Control)
Number analyzed (Participants) | 24 | 23 | 20 | 23
mL/kg/min
  Baseline | 17.9 (5.5) | 15.2 (3.2) | 15.2 (4.5) | 14.5 (4.1)
  Follow up | 19.2 (5.6) | 15.2 (3.8) | 16.5 (5.5) | 14.5 (4.1)

ADVERSE EVENTS:
Time Frame: 17 weeks
Groups:
- Aerobic Training: A customized and supervised endurance exercise training program that will last 4 months (16 weeks). The regimen will be tailored to the individual fitness level. The exercise program will consist of three supervised sessions per week. During each session, the participant will cycle on a stationary bicycle at moderate intensity for approximately 30-60 minutes.
  Exercise Training: The overall goal for all the exercise training groups will be 3 supervised exercise sessions per week an intensity between 50 to 100% of the individually determined VO2peak for aerobic training and an intensity between 50% to 85% of 1-RM for resistance training. All the exercise interventions are designed such that participants begin exercising at a low intensity (~50%-60% VO2peak / 1RM) that is subsequently increased to more moderate to vigorous intensity (~70%-100% VO2peak / ~70-85% 1RM) when appropriate. All interventions will be individually tailored to each patient following the principles of aerobic or resistance training prescription guidelines for adults.
- Resistance Training: A customized and supervised resistance exercise training program that will last 4 months (16 weeks). Resistance training will be performed on stationary weight machines, modification in equipment may be made by Exercise Physiologist. Patients will be progressively trained to perform two to three sets of 75-85% of maximal strength The participant will be trained to perform different resistance exercise, alternating between lower and upper body muscle groups. The exercise program will consist of three supervised sessions per week. Each session will last approximately 30-60 minutes.
  Exercise Training: The overall goal for all the exercise training groups will be 3 supervised exercise sessions per week an intensity between 50 to 100% of the individually determined VO2peak for aerobic training and an intensity between 50% to 85% of 1-RM for resistance training. All the exercise interventions are designed such that participants begin exercising at a low intensity (~50%-60% VO2peak / 1RM) that is subsequently increased to more moderate to vigorous intensity (~70%-100% VO2peak / ~70-85% 1RM) when appropriate. All interventions will be individually tailored to each patient following the principles of aerobic or resistance training prescription guidelines for adults.
- Combined Aerobic and Resistance Training: A customized and supervised endurance exercise training program that will last 4 months (16 weeks). The regimen will be tailored to the individual fitness level, and will be a combination of Arm A and Arm B, described above. At each session, the participant will complete aerobic training on a stationary bicycle and also resistance training using stationary weight machines. The exercise program will consist of three supervised sessions per week. Each session will last approximately 30-90 minutes.
  Exercise Training: The overall goal for all the exercise training groups will be 3 supervised exercise sessions per week an intensity between 50 to 100% of the individually determined VO2peak for aerobic training and an intensity between 50% to 85% of 1-RM for resistance training. All the exercise interventions are designed such that participants begin exercising at a low intensity (~50%-60% VO2peak / 1RM) that is subsequently increased to more moderate to vigorous intensity (~70%-100% VO2peak / ~70-85% 1RM) when appropriate. All interventions will be individually tailored to each patient following the principles of aerobic or resistance training prescription guidelines for adults.
Arm/Group | Aerobic Training | Resistance Training | Combined Aerobic and Resistance Training | Progressive Stretching Group (Attention-Control)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 8/24 | 15/23 | 12/20 | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Training (N=24) | Resistance Training (N=23) | Combined Aerobic and Resistance Training (N=20) | Progressive Stretching Group (Attention-Control) (N=23)
Abnormal heart rate response (Cardiac disorders) | 1 | 0 | 0 | 0
Abnormal blood pressure response (Vascular disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 15 | 12 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 5 | 2
Electrocardiogram abnormalities (Cardiac disorders) | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 4 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 0
Low oxygen saturation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
General fatigue (General disorders) | 2 | 5 | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5 | 4 | 0
Lower extremity fatigue (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 0
Muscle Soreness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 0
Sick (Immune system disorders) | 1 | 5 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT01068210/Prot_SAP_000.pdf